CLINICAL TRIAL: NCT00987545
Title: A Post-shave Keloid Recurrence Study in Two Parts: A Biomarker Assessment Followed by a Randomized, Double-blind, Placebo Controlled Evaluation of Safety, Tolerability, and Efficacy of QAX576
Brief Title: Efficacy 2 Part Study of Identification of Keloid Biomarkers and Effect of QAX576 on Keloid Recurrence
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Negative pharmacodynamics due to lack of Interleukin-13 signature in biomarker data from Part I of the study.
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: TKL Research, Inc. (Industry); Dermatology Consulting Services, High Point NC (Other); Skin Search (Unknown); Virginia Clinical Research, Inc. (Other)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CQAX576A2206
Record Dates: First submitted 2009-09-30; First posted 2009-10-01 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2012-05

CONDITIONS: Keloids
Keywords: Keloids; recurrence
MeSH Terms: conditions — Keloid; Recurrence

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: QAX576 placebo
- QAX576 (Experimental)
  Interventions: Drug: QAX576

INTERVENTIONS:
Drug: QAX576 — QAX576 injection
  Arms: QAX576
Drug: QAX576 placebo — Placebo to QAX576 injection
  Arms: Placebo

SUMMARY:
This is a 2-part study. In the first part (Part I, 8 subjects), biopsies will be obtained from the resection site after keloid shaving and two weeks following resection to assess and select biomarkers to determine the biologic effects that occur in shaved keloids. No drug will be administered.

In Part II (32 patients) will be randomized to receive QAX576 or placebo. An initial drug infusion will be followed by shave removal of keloids 6 - 8 days later followed by two additional drug infusions 4 weeks apart. Two weeks following resection, punch biopsies will be performed to assess biomarker responses. Patients will be followed-up for 52 weeks after first drug administration to assess keloid recurrence (clinically and by 3D imaging), and by physician's and patient's cosmetic assessments, and safety.

ELIGIBILITY:
Inclusion Criteria:

- Patients with two or more keloids on the trunk, upper extremities or thighs. The keloids must meet specified size criteria and have been present for greater than or equal to 1 year, been stable in size and symptoms for at least 6 months.

Exclusion Criteria:

* Use of other investigational drugs at the time of enrollment, or history of hypersensitivity to any of the study drugs or to drugs of similar chemical classes (e.g. lidocaine, epinephrine, and topical antibiotics as bacitracin and neomycin).
* History of repeated recurrence of keloid after prior surgical removal (4-5 times removed).
* Keloids near the hands, joints, and anogenital areas as recurrence might cause significant problems.
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of drugs, or which may jeopardize the patient in case of participation in the study

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2009-06; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Recurrence of keloids after shave removal. | At 13 weeks and 26 weeks with a follow up visit at 52 weeks after the first infusion

SECONDARY OUTCOMES:
To assess the mechanism biomarker responses post-shave removal of keloids for confirmation in Part I and application in Part II | Two weeks post-shave removal of keloids

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- United States (4):
  - TKL Research, Inc, Paramus, New Jersey
  - Skin Search of Rochester/Dermatology Associates, Rochester, New York
  - Dermatology Consulting Services, High Point, North Carolina
  - Virginia Clinical Research, Inc., Norfolk, Virginia

REFERENCES:
- See also: Results for CQAX576A2206 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=5685